CLINICAL TRIAL: NCT06303180
Title: NIDCD Otolaryngology Clinical Protocol Biospecimen Bank
Status: Recruiting | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001560; 001560-DC
Record Dates: First submitted 2024-03-08; First posted 2024-03-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11-12

CONDITIONS: Hearing Loss; Head and Neck Neoplasms; Hearing Disorders; Laryngeal Disease
Keywords: Hearing; Balance; Speech; Taste; SMELL; Tissue Sample; Genomic DNA; Saliva
MeSH Terms: conditions — Hearing Loss; Head and Neck Neoplasms; Hearing Disorders; Laryngeal Diseases; Speech

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with head and neck conditions affecting hearing, balance, smell, taste, swallowing, voice and speech.

SUMMARY:
Background:

Many disorders of the head and neck can affect a person s hearing; balance; smell; taste; swallowing; voice; or speech. These disorders include cancers and genetic and inflammatory diseases. To find better ways to diagnose and treat these disorders, researchers need to study tissues and other biological samples from people who have them.

Objective:

To collect biological samples for a repository that will be used for research.

Eligibility:

People of any age with a disorder of the head and neck that requires the taking of biological samples. The conditions may be any that affect hearing; balance; smell; taste; swallowing; voice; or speech.

Design:

Part 1: Participants will give permission for their leftover tissue samples to be used for research. These are tissue samples from the head and neck that were collected in the course of routine tests and care or other research studies. Information on each participant s age, diagnosis, and previous treatments will also be collected.

Part 2: Some participants may be asked for more samples. All those aged 3 years or older will have a physical exam. They will provide blood and saliva samples. A cotton swab or brush will be used to collect cells from the inside of the cheek.

Participants 18 years or older may have additional tests. They may provide nasal secretions: A piece of gelfoam or a sponge will be placed in the nose to soak up secretions for 5 to 10 minutes. They may have biopsies: Small samples of tissue will be cut from the skin and the tissue lining the mouth.

Samples may be used for genetic testing.

DETAILED DESCRIPTION:
Study Description:

National Institute on Deafness and Other Communication Disorders (NIDCD) investigators are studying the natural history and treatment of diverse conditions affecting hearing, balance, smell, taste, voice, speech and language at the National Institutes of Health (NIH). These studies require the collection of biospecimens for research purposes.

Objectives:

Primary:

To create a biorepository of diseased and normal tissue specimens for research purposes. The samples will be obtained:

* From surgical waste materials from participants of all ages in NIH protocols who have hearing, balance, smell, taste, voice, speech and language disorders.
* Participants aged 3 and older may have collection of blood, saliva, and/or oral swabs.
* Participants aged 18 and older, may undergo oral mucosal biopsies and skin biopsies and nasal secretion collection.

Secondary:

The specimens may be shared with other approved protocols or may be used under this protocol to conduct analysis of cellular, molecular, genetic and genomic biology of normal processes and disorders. These laboratory studies may support development of future protocols that include new therapeutic agents, novel treatment approaches, and new prognostic and diagnostic models for subjects with disorders of the head and neck affecting human communication.

Endpoints:

The primary endpoint of this study is the creation of a NIDCD biorepository from both surgical waste material and collected blood, saliva, oral swabs, nasal secretions, oral mucosa biopsy and skin biopsy specimens.

ELIGIBILITY:
* INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ability to provide their own consent, or for minors, a parent or guardian is able to consent on their behalf.
* Ability of subject (or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Have a hearing, balance, smell, taste, voice, speech or language condition for which the subject is under clinical care or research purposes under a separate Review Board (IRB) approved protocol; OR be a healthy volunteer aged at least 3 years, enrolled on an approved research protocol.

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

* Have active symptomatic major organ disorders that would increase the risk of biopsy for research, including but not limited to bleeding disorders, ischemic heart disease, a recent myocardial infarction, active congestive heart failure or severe pulmonary dysfunction
* Have specific medical condition, such as a bleeding tendency where additional biopsies or phlebotomy procedures may increase the subjects risk in participating. This will be determined at the discretion of the principal investigator.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 subjects of any age, any race, ethnicity and gender. Only viable neonates will be enrolled. We are hoping to accrue about 100 subjects a year over 10 years. NIH employees and staff participating in an approved NIH protocol. There will be no collection or recruitment of healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2033-12-30 (Estimated); Study Completion 2033-12-30 (Estimated)

PRIMARY OUTCOMES:
To create a biorepository of diseased and normal tissue specimens for research purposes. | Ongoing
  (Part 1) From surgical waste materials from participants of all ages in NIH protocols who have head and neck disorders.(Part 2) Participants aged 3 and older may have collection of blood, saliva, and/or oral swabs. Participants aged 18 and older, may undergo oral mucosal biopsies and skin biopsies and nasal secretion collection, taken from subjects with head and neck disorders.

SECONDARY OUTCOMES:
To share specimens with the NCI Frederick Patient-Derived Xenograft (PDX) team, other approved protocols or may be used under this protocol to conduct analysis of cellular, molecular, genetic and genomic biology of | Ongoing
  These laboratory studies may support development of future protocols that include new therapeutic agents, novel treatment approaches, and new prognostic and diagnostic models for subjects with disorders of the head and neck affecting human communication

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Levy, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001560-DC.html